CLINICAL TRIAL: NCT05456009
Title: Exhaled Breath Analysis by Secondary Electrospray Ionization - Mass Spectrometry (SESI-MS) in Human Subjects
Brief Title: Exhaled Breath Analysis in Human Subjects
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Deep Breath Intelligence (DBI) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-00030
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Exhaled Breath Pattern After Medication Intake, in OSA Patients, or Other Pulmonary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Identification of exhaled breath pattern of human subjects

DETAILED DESCRIPTION:
Breath analysis with mass spectormetry as a non-invasive method to identfy exhaled breath patterns.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years
* Informed consent

Exclusion Criteria:

* specific exclusion criteria for different subgroups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of human subjects with heart failure, dementia syndrome, parkinson disease, obstructive sleep apnea, chronic obstructive pulmonary disease, pneumonia, specific medication use.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Exhaled breath pattern | baseline
  mass spectrometric profile of exhaled breath pattern of human subjects

SECONDARY OUTCOMES:
Chemical structure of exhaled breath molecules | baseline
  The identification of the chemical structure of exhaled breath molecules
Body fluids | baseline
  The correlations of identified molecules in exhaled breath with body fluids
Disease marker | baseline
  The correlation of a distinct disease marker with a breath print or breath feature
Distinguish between disease | baseline
  The use of a breath print to distinguish between disease and/or health state
Health state | baseline
  The correlation of breath prints to subjective health state and/or quality of life
Medication | baseline
  Response to medication and toxicity as a function of blood/breath drug concentrations
Excretion of drugs | baseline
  Correlation between lung function and the excretion of drugs in exhaled breath

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
if requested